CLINICAL TRIAL: NCT03561493
Title: Effect of Zumba Exercise on Menstrual Pain in Women With Primary Dysmenorrhea
Brief Title: The Effect of Zumba Dance on Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zumba exercise
Record Dates: First submitted 2018-05-11; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zumba exercise group (Experimental): Participants will engage in 16 classes of 60-minute Zumba® fitness for two consecutive menstrual cycles (an 8-week period, twice weekly). Each class was one h in length and a recovery period of at least 48 h was taken between classes.
  Interventions: Other: zumba exercise
- non zumba exercise group (No Intervention): The participants in the control group did not receive any intervention.

INTERVENTIONS:
Other: zumba exercise — Participants will engage in 16 classes of 60-minute Zumba® fitness for two consecutive menstrual cycles (an 8-week period, twice weekly). Each class was one hour in length and a recovery period of at least 48 h was taken between classes. Each session will be initiated with low-intensity movements for the ﬁrst 5 min, followed by an increasing intensity throughout the workout. At the end of the training session, the intensity will be gradually reduced. The Zumba sessions will be supervised by three certiﬁed Zumba instructors, each responsible for regular sessions per week.
  Other Names: zumba fittness
  Arms: zumba exercise group

SUMMARY:
the objective of this study is to investigate the effect of practising Zumba exercise in decreasing menstrual pain in young women with primary dysmenorrhea.

DETAILED DESCRIPTION:
primary dysmenorrhea or painful menstruation without pelvic pathology is one of the most common complaints in women's medicine. The pain begins with the onset of menstrual bleeding and lasts for 72-12 h. Pain is usually in the middle line of the highest severity. Dysmenorrhea pain is often described as cramped and intermittent. Zumba is a dance-based fitness class that originated in Colombia in the 1990s and is now extremely popular worldwide. the aim of this study is to investigate the effect of 8 weeks of regular Zumba exercise on the severity of primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* having regular menstrual cycles (30-35 days) and bleeding time of 3-10 days.
* history of primary dysmenorrhea(PD) which had affected daily activities in at least 50% of their cycles through the past 6 months; and pain intensity over 4 cm, based on the 10-cm visual analog scale score.
* having a pain score for PD on the visual analog scale (VAS) of 4-7 cm
* Age: 18-25 years.

Exclusion Criteria:

* Pregnancy
* known diseases of the genitourinary system (e.g., pelvic inflammatory disease and urinary tract infections) or secondary dysmenorrhea and chronic diseases (heart disease, respiratory, kidney, blood pressure, asthma, diabetes, epilepsy, migraine, thyroid, anemia, nervous disorders).
* Previous Zumba fitness practice.
* irregular menstrual cycles; the use of intra-uterine devices and oral contraceptive pills.
* musculoskeletal injuries and metabolic/cardiorespiratory contraindications to physical exercise

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-06-25 (Estimated); Primary Completion 2018-09-25 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Intensity of pain | duration of menses(5-7 days) 1st menstrual cycle.
  Pain intensity will be measured by using a 10-point visual analog scale(VAS) in which a line was calibrated from 0 to 10 with 0 representing ''no pain at all''and 10 representing ''worst pain possible.'' Participants will indicate their perceived pain levels by pointing to the appropriate value on a 10-cm horizontal ruler. The intensity of pain will be rated to the ﬁrst decimal place in centimeters.Higher scores represent higher menstrual pain intensity.
Intensity of pain | duration of menses(5-7 days) 2nd menstrual cycle.
  Pain intensity will be measured by using a 10-point visual analog scale(VAS) in which a line was calibrated from 0 to 10 with 0 representing ''no pain at all''and 10 representing ''worst pain possible.'' Participants will indicate their perceived pain levels by pointing to the appropriate value on a 10-cm horizontal ruler. The intensity of pain will be rated to the ﬁrst decimal place in centimeters.Higher scores represent higher menstrual pain intensity.

SECONDARY OUTCOMES:
menstrual pain duration | 7 days from 1st day of menstruation).
  duration of menstrual pain in days will be measured by using descriptive data that will be obtained from study participants.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University